CLINICAL TRIAL: NCT00062296
Title: Phase II Study of Epirubicin and Rituximab in Relapsed and Refractory B-Cell Non-Hodgkin's Lymphoma and CLL
Brief Title: Epirubicin and Rituximab in Treating Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: FCCC-02025; CDR0000304711 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: rituximab
Drug: epirubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as epirubicin use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining epirubicin with rituximab may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining epirubicin with rituximab in treating patients who have relapsed or refractory B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, time to progression, and overall survival of patients with refractory or relapsed B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia treated with epirubicin and rituximab.
* Determine the toxicity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a non-randomized, open-label, multicenter study.

Patients receive epirubicin IV over 3-5 minutes once weekly for 6 weeks. Patients also receive rituximab IV on weeks 2 and 5 during course 1 and then on weeks 1 and 4 for all remaining courses. Treatment repeats every 8 weeks for a maximum of 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 18-38 patients will be accrued for this study within 2.5-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed B-cell non-Hodgkin's lymphoma (any grade) or chronic lymphocytic leukemia meeting 1 of the following criteria:

  * Primary refractory disease
  * Disease progression after at least 1 but no more than 4 prior cytotoxic chemotherapy regimens

    * Rituximab administered alone is not considered 1 prior regimen
    * High-dose chemotherapy with stem cell support is considered 1 prior regimen
* Bidimensionally measurable or evaluable disease outside prior irradiation port
* No clinical evidence of CNS involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 2,000/mm^3*
* Platelet count at least 100,000/mm^3* NOTE: *Unless due to bone marrow involvement

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT no greater than 2 times upper limit of normal (ULN)

Renal

* Creatinine no greater than 2 times ULN

Cardiovascular

* No unstable angina
* No uncontrolled congestive heart failure
* LVEF at least 45%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study treatment
* HIV negative
* No other concurrent primary malignancy except basal cell or squamous cell skin cancer, carcinoma in situ, or localized solid tumors cured more than 5 years ago
* No acute infection requiring systemic therapy
* No confusion, disorientation, or major psychiatric illness that would preclude understanding of informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 4 weeks since prior biologic therapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* Prior cumulative doxorubicin dose no greater than 6 courses at 50 mg/m^2

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to the entire pelvis
* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 7 days since prior cimetidine
* No concurrent cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R. Smith, MD, PhD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States